CLINICAL TRIAL: NCT01098071
Title: Open Label Pilot Trial, Evaluating the Role of Nasonex in the Management of Nasal Obstruction Secondary to Adenoids Hypertrophy in Children
Brief Title: Nasonex (Mometasone Furoate Nasal Spray) in Adenoids Hypertrophy in Children (P04367)
Acronym: NAHCh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04367 - Lebanon
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Adenoids
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mometasone furoate nasal spray (Experimental)
  Interventions: Drug: mometasone furoate nasal spray

INTERVENTIONS:
Drug: mometasone furoate nasal spray — One spray (50 mcg per spray) in each nostril once daily (100 mcg daily) for 3 months
  Other Names: SCH 32088; Nasonex

SUMMARY:
To document the short term & long term effect of treatment with Nasonex (mometasone furoate nasal spray) in moderate to severe adenoids hypertrophy (which cause > 50% obstruction of the posterior choanae).

ELIGIBILITY:
Inclusion Criteria:

* 2-11 years of age, nasal obstruction for 3 months, adenoids hypertrophy > 50% of posterior choanae.

Exclusion Criteria:

* adenoids hypertrophy < 50% of posterior choanae

recurrent epistaxis or immunodeficiency, severe septal deviation, kissing tonsils, choanal atresia, large masses, known allergy to nasonex (mometasone furoate nasal spray), chronic otitis media, cystic fibrosis, acute infection.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2009-09-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bitar MA, Mahfoud L, Nassar J, Dana R. Exploring the characteristics of children with obstructive adenoid responding to mometasone fuorate monohydrate: preliminary results. Eur Arch Otorhinolaryngol. 2013 Mar;270(3):931-7. doi: 10.1007/s00405-012-2155-8. Epub 2012 Aug 22. PMID 23010795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray
Started | 34
Completed | 19
Not Completed | 15
Not completed — Surgery (adenoidectomy) | 2
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 34
Age, Customized [Mean (Full Range); unit: Years] | 4.84 [0.5 to 9.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Region of Enrollment [Number; unit: participants]
  Lebanon | 34

OUTCOME MEASURES:

1. Primary Outcome: Severity of Nasal Obstruction Symptoms at Baseline and Week 12 as Measured by the Total Clinical Score
Description: Clinical score (based on a 5 point grading system) was assessed for each of 5 nasal obstruction symptoms (oral/mouth breathing, snoring, restless sleep, frequent waking-ups during the night, and obstructive breathing during sleep). Each nasal obstruction symptom was estimated by the parent/guardian of the participant and scored on a scale of 0 (best) to 1 (worst). Total clinical score is a score on a scale (0 = no symptoms [best score] and 5 = worst symptoms [worst score]).
Time Frame: Baseline and Week 12
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 19
Score on a scale
  Baseline score | 3.89 [2 to 5]
  Score at Week 12 | 1.26 [0 to 4]

2. Primary Outcome: Degree of Posterior Choana Obstruction at Baseline and Week 12
Description: The degree of obstruction of the posterior choana was assessed by endoscopy. Endoscopy grading consisted of Grade I (minimum), Grade II and Grade III (maximum). Grade I was defined as <50% obstruction, Grade II was defined as 50-75% obstruction, and Grade III was defined as >75% obstruction.
Time Frame: Baseline and Week 12
Population: Only participants that completed the study are included.
Measure: Mean (Full Range); unit: Percent obstruction
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 19
Percent obstruction
  Baseline score | 85 [70 to 90]
  Score at Week 12 | 61 [40 to 80]

3. Primary Outcome: Number of Participants Referred to Surgery (Adenoidectomy) Within 12 Weeks of Start of Therapy
Time Frame: Baseline to 12 weeks
Population: Evaluable population (per protocol population, ie, those participants without protocol violation of inclusion or exclusion criteria)
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 19
Participants | 2

4. Secondary Outcome: Severity of Rhinorrhea at Baseline and Week 12
Description: Rhinorrhea is a symptom of allergic rhinitis. Rhinorrhea was assessed using a 3-point scale (0 = no symptoms [best score] and 3 = symptom interferes with daily life activity [worst score]).
Time Frame: Baseline and Week 12
Population: Participants suspected to have allergic rhinitis
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 10
Score on a scale
  Baseline score | 0.95 [0 to 3]
  Score at Week 12 | 0.37 [0 to 2]

5. Secondary Outcome: Severity of Nasal Congestion at Baseline and Week 12
Description: Nasal congestion is a symptom of allergic rhinitis. Nasal congestion was assessed using a 3-point scale (0 = no symptoms [best score] and 3 = symptom interferes with daily life activity [worst score]).
Time Frame: Baseline and Week 12
Population: Participants suspected to have allergic rhinitis
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 10
Score on a scale
  Baseline score | 0.79 [0 to 3]
  Score at Week 12 | 0.32 [0 to 3]

6. Secondary Outcome: Severity of Nasal Itching at Baseline and Week 12
Description: Nasal itching is a symptom of allergic rhinitis. Nasal itching was assessed using a 3-point scale (0 = no symptoms [best score] and 3 = symptom interferes with daily life activity [worst score]).
Time Frame: Baseline and Week 12
Population: Participants suspected to have allergic rhinitis
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 10
Score on a scale
  Baseline score | 0.74 [0 to 3]
  Score at Week 12 | 0.37 [0 to 1]

7. Secondary Outcome: Severity of Sneezing at Baseline and Week 12
Description: Sneezing is a symptom of allergic rhinitis. Sneezing was assessed using a 3-point scale (0 = no symptoms [best score] and 3 = symptom interferes with daily life activity [worst score]).
Time Frame: Baseline and Week 12
Population: Participants suspected to have allergic rhinitis
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 10
Score on a scale
  Baseline score | 0.89 [0 to 3]
  Score at Week 12 | 0.37 [0 to 2]

8. Secondary Outcome: Severity of Eye Symptoms at Baseline and Week 12
Description: Eye symptoms are a symptom of allergic rhinitis. Eye symptoms were assessed using a 3-point scale (0 = no symptoms [best score] and 3 = symptom interferes with daily life activity [worst score]).
Time Frame: Baseline and Week 12
Population: Participants suspected to have allergic rhinitis
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 10
Score on a scale
  Baseline score | 0.68 [0 to 3]
  Score at Week 12 | 0.16 [0 to 1]

ADVERSE EVENTS:
Description: In this study, symptoms of allergic rhinitis (rhinorrhea, nasal congestion, nasal itching, sneezing, and eye symptoms) were not reported as adverse events.
Arm/Group | Mometasone Furoate Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator and his co-workers agree not to publish or publicly present any results of the study without the prior written consent and approval of the sponsor.